CLINICAL TRIAL: NCT01986777
Title: LDX in the Treatment of Executive Function Difficulties in Women After Oophorectomy
Brief Title: LDX for the Treatment of Cognitive Functioning Issues in Women Post-Oophorectomy
Acronym: LDX
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not obtained
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 817628
Record Dates: First submitted 2013-10-30; First posted 2013-11-18 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Cognitive Impairments; RRSO
Keywords: cognitive complains; RRSO; oophorectomy; memory; cognition; early menopause
MeSH Terms: conditions — Cognitive Dysfunction; Primary Ovarian Insufficiency | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- lisdexamfetamine (Active Comparator): Participants will have a 50% chance of receiving the active study medication. They will begin at 20 mg/d and will increase up to 60 mg/d after 4 weeks, if well tolerated. Total time on the study drug is up to 10 weeks.
  Interventions: Drug: lisdexamfetamine
- Placebo (Placebo Comparator): Participants will have a 50% chance of receiving the placebo for this study. They will begin with 1 sugar pill and will increase up to 3 pills after 4 weeks. Maximum time for taking the placebo is 8-10 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lisdexamfetamine
  Other Names: Vyvanse
  Arms: lisdexamfetamine
Drug: Placebo — The placebo capsules will be filled with lactose.
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled, study testing whether LDX improves cognitive function and EF in 20 postmenopausal women who report onset of cognitive difficulties after oophorectomy (with or without subsequent chemo/adjunctive therapy). Brain imaging is included at critical time points to obtain objective data regarding effects of LDX as well as potential predictors of resilience in the face of oophorectomy.

DETAILED DESCRIPTION:
Participants will be asked to undergo three brain-imaging scans throughout the course of the study. Once they are deemed eligible for participation based on two assessment visits, they will be scheduled for their baseline test day. On this they, they will be asked to under a series of cognitive tests following by a brain-imaging scan. They will then take the first dose of either the LDX or placebo, wait for 3 hours and then undergo another brain-imaging scan to assess acute changes to memory/cognition due to the study drug. They will then come in for three 30-minute check-in visits during weeks 2, 4 and 6 on the study drug. They will be asked to undergo a final scan and series of cognitive tasks during weeks 8-10 on the study drug. They will then be discharged from active study participation. All participants, regardless of randomization, will be offered a consultation with the study MD and optional prescription for 4-weeks of treatment with LDX.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Age 30-60;
* Have undergone surgically-induced menopause by oophorectomy or chemically-induced menopause within the previous 10 years;
* Have at least moderate executive functioning difficulties as evidenced by a score of 25 on the BADDS;
* Have no history of a DSM-IV psychiatric disorder within the previous year or substance dependence disorder within the previous 5 years (psychostimulant abuse lifetime history), according to the Structured Clinical Interview for Diagnosis-DSM-IV (SCID)-Non-Patient Version;
* Subject has history of substance abuse disorders (this includes alcohol, prescription, and illicit substances) 3 years ago but the period of abuse did not last more than 5 years according to the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-NP);
* Are able to give written informed consent (obtained at screening visit);
* Must have clear urine toxicology screen upon recruitment;
* Are fluent in written and spoken English;
* Are right-handed.

Exclusion Criteria:

* Mini-mental status exam score of 24;
* Presence of a psychiatric disorder within previous year or a life time history of ADHD or psychotic disorder including bipolar disorder, schizoaffective disorder and schizophrenia;
* Lifetime history of drug addiction or abuse, except nicotine; 4. Regular use of psychotropic medication except for a selective serotonin reuptake inhibitor or serotonin/norepinephrine reuptake inhibitor or standard sleep medication at a stable dose for at least one month prior to enrollment;
* Regular use (more than once a week) of alcohol that is 3 drinks/day;
* Presence of a contraindication to treatment with stimulant medication; this would include the presence of controlled or uncontrolled hypertension, coronary disease, atrial fibrillation, and arrhythmia;
* History of seizures;
* History of cardiac disease including known cardiac defect or conduction abnormality;
* Abnormal electrocardiogram during screening;
* Presence of a metallic implant;
* Claustrophobia.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
BADDS Score | 8-10 weeks
  To determine whether treatment with LDX improves self-reported executive function (EF) as measured with the BADDS

SECONDARY OUTCOMES:
Brain Activation | 8-10 weeks
  To determine the impact of LDX on brain activation in the brain during a working memory task.

CONTACTS AND LOCATIONS:
Overall Officials: C. Neill Epperson, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Center for Women's Behavioral Wellness, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Study has been withdrawn